CLINICAL TRIAL: NCT06373965
Title: An Online HIV Self-testing Intervention with Online-to-offline Linkage to Care for Transgender Women
Brief Title: Integrated Online-to-offline (O2O) Model of Care for HIV Prevention and Treatment Among Transgender Women (CINTAI)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: University of Malaya (Other)
Responsible Party: Principal Investigator, Roman Shrestha, Assistant Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B2024-000
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: HIV Prevention Program
Keywords: HIV; transgender women

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CINTAI (Experimental): Participants randomized to the Jom-TestPlus group will have access to all Jom-TestPlus features, including: assessment center; online registration; risk calculator; HIVST kit order, management, and monitoring; automated reminders; real-time e-counseling (eHIVST, active referral services); chemsex-related harm reduction services (screening, chemsex e-counseling, PartyPack ordering), chat function (ability to chat with counselors and research staff); and knowledge center (multimedia library on information and resources on HIV testing, PrEP, treatment, risks, and chemsex). Participants will follow a defined pathway to accessing HIVST kit ordering, e-counseling, and subsequent O2O linkage to clinical services.
  Interventions: Behavioral: Online to offline counseling
- Control (Active Comparator): The TAU group will have access to the assessment center (risk assessment, follow-up surveys), knowledge center (multimedia library on information and resources on HIV testing, PrEP, treatment, risks, and chemsex), and a voucher for no-cost community-based HIV testing (sent via secure, encrypted email or can be downloaded on the Jom-TestPlus).
  Interventions: Behavioral: Online to offline counseling

INTERVENTIONS:
Behavioral: Online to offline counseling — * Online registration and risk assessment: Users complete an onboarding process comprised of creating an account, entering demographic data, customizing settings, and completing the baseline risk assessment.
  * HIVST kit order, management, and monitoring: The platform will allow users to request HIVST kits via standard mail or self-pickup at user-preferred sites (e.g., LGBT-friendly clinics). After completing the mandatory section of the questionnaire and selecting a delivery option, a random personal identification number will be assigned by the system, which will be used to track future HIVST requests, collect HIVST results, and monitor subsequent linkage to further testing and HIV care.
  * eHIVST and O2O linkage to HIV clinical services: After unsealing the test kit, participants will find a reminder card to schedule their O2O pre- and post-test e-counseling appointment.

SUMMARY:
The proposed research focuses on developing and testing a web-based platform, called Jom-TestPlus, that will incorporate HIV self-testing (HIVST) with real-time e-counseling (eHIVST) with online-to-offline (O2O) linkage to HIV prevention and treatment services while simultaneously co-addressing chemsex-related needs for transgender women (TGW) in Malaysia. This model represents a potentially impactful strategy for reaching marginalized populations, like TGW, and allows immediate engagement in the post-test linkage process to prevention or treatment services.

DETAILED DESCRIPTION:
Globally, transgender women (TGW) are disproportionately impacted by the HIV epidemic, with an estimated HIV prevalence of 19.1%. Malaysia, one of SE Asia's fastest-growing economies, is witnessing a rapid transition to its HIV epidemic. Malaysia has an estimated 80,000 TGW in-country, of which 12.4% are living with HIV. TGW experience numerous unique vulnerabilities to HIV, including discrimination in employment and economic opportunities, steering many TGW into high-risk occupations, such as sex work. High levels of stigma and discrimination against TGW by healthcare providers can foster a hostile environment toward TGW, complicating efforts to scale-up of HIV testing and prevention services among trans women, including preexposure prophylaxis (PrEP). Modeling studies suggest that increased HIV testing and uptake of PrEP is the most impactful and cost-effective strategy for reducing new infections. Despite this, only 37% of TGW in Malaysia have ever been HIV tested. HIV self-testing (HIVST) may be particularly impactful among TGW in Malaysia, where anti-trans stigma persists. Although willingness to use HIVST is high (48%) among Malaysian TGW, its use is still minimal due to a lack of access to HIVST kits, concerns related to misinterpreting results, and missed opportunities for counseling and linkage to care. In this context, eHealth represents an innovative platform to transform the face of HIV service delivery (i.e., HIVST and linkage to care). Leveraging eHealth technology for HIV services delivery is ideal given that nearly all (>93.6%) TGW use online technology (e.g., smartphone, tablet, computer) and indicate a strong preference for a web-based platform for HIVST. As such, HIVST with real-time e-counseling (eHIVST), integrated with online-to-offline (O2O) linkage to prevention and treatment, offers an innovative and empowering approach that could transform TGW's uptake of HIV testing and engagement in the broader HIV care continuum. This proposal - submitted in response to the Notice of Special Interest (Administrative Supplements for Research on Sexual and Gender Minority Populations; NOT-OD-22-032) - requests an SGM administrative supplement to add a sample of TGW to parent award (R34MH130233), a project that focuses on developing and testing a web-based platform, called Jom-TestPlus, that will incorporate an O2O service delivery model with eHIVST that facilitates rapid linkage to the HIV prevention and treatment continuum for men who have sex with men (MSM) in Malaysia. Expanding Jom-TestPlus to include TGW represents a significant opportunity to leverage existing resources from the parent award to address HIV and other health inequities among broader SGM populations. If successful, Jom-TestPlus will serve as a model that can easily be adapted for various health outcomes and healthcare services delivery in these populations and other LMICs.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Cisgender male;
* HIV-negative or HIV status unknown;
* Own or have access to a computer, tablet, or internet-enabled smartphone

Exclusion Criteria:

* Currently on PrEP
* Unable to provide informed consent
* Unable to read and understand English or Bahasa Malaysia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-08-13 (Actual); Primary Completion 2025-12-06 (Estimated); Study Completion 2026-12-18 (Estimated)

PRIMARY OUTCOMES:
HIVST uptake | Time Frame: 3 and 6 months post-randomization
  Uptake of HIV self-testing (yes/no) will be assessed at each follow-up time point (3 and 6 months) using self-reported measure.
Linkage to PrEP | Time Frame: 3 and 6 months post-randomization
  Linked to PrEP (yes/no) will be assessed at each follow-up time point (3 and 6 months) using self-reported measure.
Linkage to HIV treatment services | Time Frame: 3 and 6 months post-randomization
  Linked to ART services (yes/no) will be assessed at each follow-up time point (3 and 6 months) using self-reported measure.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre of Excellence for Research in Infectious Diseases and AIDS (CERiA), University Malaya, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No